CLINICAL TRIAL: NCT05360316
Title: The Effect of Extracorporeal Shock Wave Therapy Applied to the Plantar Region in Individuals With Hemiplegia on Mobility, Plantar Pressure Distribution and Sensory
Brief Title: Extracorporeal Shock Wave Therapy Applied to the Plantar Region in Individuals With Hemiplegia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Furkan BİLEK, Principal Investigator, Firat University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Firat Uni
Record Dates: First submitted 2022-04-16; First posted 2022-05-04 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Extracorporeal Shock Wave Therapy; Kinaesthesia; Sensory Disorders
Keywords: Extracorporeal Shock Wave Therapy; Kineaesthesia; Hemiplegia; Deep sense; Superficial sense
MeSH Terms: conditions — Sensation Disorders; Hemiplegia

STUDY DESIGN:
Intervention Model Description: randomized controlled, double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESWT (Placebo Comparator): Patients assigned to the ESWT group received ESWT over the plantar fascia, three days/week, for six weeks. In addition patients participated additional in the same conventional stroke rehabilitation program consisting of 60 minutes of treatment a day, five times a week for six weeks (30 sessions). The conventional therapy programs were patient-specific and consisted mainly of physiotherapy, such as neurodevelopmental facilitation techniques, passive mobilization, occupational therapy, postural control exercises, stretching and range-of-motion exercises for the hemiparetic side and balance training.
  Interventions: Device: ESWT
- Placebo (No Intervention): Routine therapy Patients participated in the same conventional stroke rehabilitation program consisting of 60 minutes of treatment a day, five times a week for six weeks (30 sessions). The conventional therapy programs were patient-specific and consisted mainly of physiotherapy, such as neurodevelopmental facilitation techniques, passive mobilization, occupational therapy, postural control exercises, stretching and range-of-motion exercises for the hemiparetic side and balance training.

INTERVENTIONS:
Device: ESWT — extracorporeal shock wave therapy
  Arms: ESWT

SUMMARY:
Sensory and balance losses occur in hemiplegic patients. In some patients, sensory and balance rehabilitations may vary depending on the treatment they receive, depending on the treatment. It is a fact that the affected anatomic neuronal regions can cause different damages for each person together with interneuronal relations. This study aims to sense sensation with Extracorporeal Shock Wave Therapy to be applied to the plantar region.

DETAILED DESCRIPTION:
Every year in England and Wales, 110,000 people experience first stroke and 30,000 people experience other stroke events following the first stroke. Stroke is one of the most important events causing severe distress and is shown as the third most common cause of death in England. Most of the health and social care resources budget uses it to meet the acute and chronic care of stroke patients. 5% of all hospital expenses are spent for the care of stroke patients. Stroke causes 88% of the death causes of the 65 and over life group and 10-12% of all deaths in industrial countries. Stroke can always be an obstacle in patients and cause them to need long-term care. After the stroke, patients apply to the hospital due to psychological, social and physical problems. The sudden loss of functionality creates strong stress not only in the patient but also in the family. Neurological damage can also become irreversible distress. Signs and symptoms related to stroke vary depending on the localization and severity of the damage. Stroke often results in paralysis of one side of the body. Paralysis of one side of the body occurs on the opposite side of the damaged side of the brain. Stopping blood flow to the brain causes focal function loss up to various levels in the patient. The most common motor is loss. Other neurological losses are visual, sensory, communicative, swallowing and perceptual problems.

Kinesthesis and vibration losses are especially evident in the distal parts of the extremities. Kinesthesis and loss of position sense cause irregular and excessively flawed movements that are performed voluntarily with insufficient information about proprioception to the sensory cortex. Such patients are able to stand or walk, although they are not very balanced, as they can somewhat assess the position of their body parts with the sense of vision; but they have great difficulty walking in the dark.

Shock waves have been used extensively to study their effects on sensory nerves and nerve endings. Application of 1000 impulses of shock waves (0.08 mJ/mm, 2.4 Hz) resulted in the degeneration of sensory nerve fibers and endings followed by reinnervation of the affected skin areas These changes were accompanied by the reversible and rapid loss of the immunohistochemical markers protein gene product 9.5 and calcitonin gene-related peptide. However, a second application of the same dose of shock waves had a cumulative effect on the treated nerves, leading to delayed reinnervation. It appears, therefore, that shock wave-treated nerves develop a "memory effect" after the first treatment, and Extracorporeal Shock Wave Therapy (ESWT) repeated shortly after the first treatment is not beneficial. It is expected that ESWT induces subtle changes in the affected neurons whose axons have been treated. Investigators detected an increased expression of activating transcription factor 3 (ATF-3) and growth-associated phosphoprotein 43 (GAP-43) in dorsal root ganglion neurons of shock wave-treated rats, indicating that the molecular changes after ESWT are not restricted to the treated axons: their cell bodies are also activated in a retrograde manner. The question remains open as to whether doses of ESWT in the therapeutic range would induce similar changes as the 2000 impulses applied in this study. ATF-3 and GAP-43 are markers thought to be associated with the activation of neurons and glial cells (Schwann cells) after peripheral nerve injuries.

As regards the dose-effect relationship of ESWT on peripheral nerves, a large body of evidence suggests that shock wave doses greater than 900 impulses combined with a flux density of 0.08 mJ/mm2 induce damage to the affected nerves, manifested in impaired electrophysiological conduction parameters, a disrupted neurofilament staining pattern of the treated axons, and degeneration of the myelin sheaths at the levels of light and electron microscopy. These doses appeared to damage motor and sensory nerves equally. This experimental and clinical experience indicates that the therapeutically applicable dose for the promotion of nerve regeneration without side effects is likely to be lower than 500 impulses. The effect of such doses is highly dependent on the depth of the target tissue and the treated surface area.

In this study, the effect of ESWT on sensory nerves will be used in individuals with hemiplegia. Thus, mobility and plantar region sensory development of plantar sensory stimulation will be evaluated in individuals with hemiplegia. A study specific to the literature will be presented by evaluating the effect of evaluation results on the function.

ELIGIBILITY:
Inclusion Criteria:

* First-ever hemiplegia
* Hemiplegia duration of at least 6 months
* Ability to walk alone without an orthosis.

Exclusion Criteria:

* Patients with ataxia, dystonia, or dyskinesia
* Patients with dementia
* Patients with bilateral hemiplegia
* Taking antispastic drugs

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-04 (Actual); Primary Completion 2021-04-04 (Actual); Study Completion 2021-05-04 (Actual)

PRIMARY OUTCOMES:
Balance | 3 mounths
  Berg Balance Scale (BBS): The BBS is a 14-item test of functional balance, with each item rated out of 4 for a total score of 56. It assesses static balance in sitting and standing, as well as dynamic balance during transitions and while in standing. Individuals who are able to maintain their balance for each task score higher on this outcome.
Maximum plantar pressure | 3 Mounths
  The Win-Track platform (MEDICAPTEURS Technology, France) is a tool used to measure maximum plantar pressure
Static posture | 3 Mounths
  The Win-Track platform (MEDICAPTEURS Technology, France) is a tool used to measure static posture
Step cycle duration | 3 Mounths
  The Win-Track platform (MEDICAPTEURS Technology, France) is a tool used to measure step cycle duration
Single-support phase | 3 Mounths
  The Win-Track platform (MEDICAPTEURS Technology, France) is a tool used to measure single-support phase
Swing phase | 3 Mounths
  The Win-Track platform (MEDICAPTEURS Technology, France) is a tool used to measure swing phase
Step length | 3 Mounths
  The Win-Track platform (MEDICAPTEURS Technology, France) is a tool used to measure step length
Foot angle | 3 Mounths
  The Win-Track platform (MEDICAPTEURS Technology, France) is a tool used to measure foot angle
Cadence | 3 Mounths
  The Win-Track platform (MEDICAPTEURS Technology, France) is a tool used to measure cadence
Gait cycle distance | 3 Mounths
  The Win-Track platform (MEDICAPTEURS Technology, France) is a tool used to measure

CONTACTS AND LOCATIONS:
Overall Officials: Gulnihal Deniz, Asst. Prof., Study Chair — Firat University
Locations (1):
- Furkan Bilek, Elâzığ, Turkey (Türkiye)